CLINICAL TRIAL: NCT00797459
Title: A Randomized, Double-Blind Study Comparing Safety and Tolerability of Restylane® With and Without Addition of 0.3% Lidocaine HCL During Correction of Nasolabial Folds
Brief Title: Safety & Tolerability Study That Compares Restylane to Restylane With Lidocaine While Correcting Wrinkles in the Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Collaborators: Q-Med Scandinavia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MA-1100-001
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Nasolabial Folds
Keywords: Correction of Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane and Restylane with Lidocaine (Experimental): This is a split-face design injecting both Restylane and Restylane-L injectable gels, administered once. Each subject received Restylane on one side of the face, and Restylane-L on the other. Subjects were blinded to which side of their face received Restylane or Restylane-L. The study was randomized and treatments successive.
  Interventions: Device: Restylane and Restylane-L

INTERVENTIONS:
Device: Restylane and Restylane-L — This is a split face design and each subject received both Restylane and Restylane-L. Treatments were double blind, randomized, and successive.

SUMMARY:
Safety & tolerability study that compares Restylane to Restylane with Lidocaine (Restylane-L) while correcting wrinkles in the area around your nose.

DETAILED DESCRIPTION:
A Randomized, Double-Blind Study Comparing Safety and Tolerability of Restylane® With and Without Addition of 0.3% Lidocaine HCL During Correction of Nasolabial Folds

ELIGIBILITY:
Inclusion Criteria:

* Subjects seeking augmentation therapy for correction of bilateral NLFs
* Same WSRS score at both NLFs (either both Moderate [3] or both Severe [4])
* Subjects willing to give written informed consent to participate in the study
* Women of childbearing potential willing to use an acceptable form of birth control during the study period

Exclusion Criteria:

* Active or chronic skin disease, inflammation or related conditions, near or on the NLFs
* Subjects who had undergone procedures based on active dermal response e.g., laser or chemical peeling procedures) within 6 months prior to study entry
* Use of any facial tissue augmenting therapy with non-permanent filler or aesthetic facial surgical therapy within 9 months prior to study entry
* Permanent implant placed in the NLF area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bank, MD, Principal Investigator — The Center for Dermatology, Cosmetic and Laser Surgery; Fredric Brandt, MD, Principal Investigator — Dermatology Research Institute LLC; Robert Weiss, MD, Principal Investigator — Maryland Laser Skin and Vein Institute; Ron Staugaard, Study Director — Medicis Pharmaceutical
Locations (3):
- United States (3):
  - Dermatology Research Institute LLC, Coral Gables, Florida
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland
  - The Center for Dermatology, Cosmetic and Laser Surgery, Mount Kisco, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Restylane: Split-face design with each subject receiving Restylane on one side of the face and Restylane with Lidocaine (Restylane-L) on the other. Injection frequency is once on day 1.
Period: Overall Study
Arm/Group | Restylane
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Restylane
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Treatment Difference in Pain as Measured by a Visual Analogue Scale
Description: No pain is noted at 0 mm and worst pain is noted at 100 mm.
Time Frame: After Injection on Day of Treatment
Population: This is a split-face design. Restylane and Restylane with Lidocaine was injected to different sides of the subject's face. A total of 60 subjects received both products. The study evaluated which side of the face had less pain, as measured by the Visual Analogue Scale (VAS).
Measure: Mean (Standard Deviation); unit: Scores on a VAS Scale
Units Other Than Participants: Scores on a Scale
Groups:
- Restylane-L: Split-face design with each subject receiving Restylane on one side of the face and Restylane with Lidocaine (Restylane-L) on the other. Injection frequency is once on day 1.
Arm/Group | Restylane | Restylane-L
Number analyzed (Participants) | 60 | 60
Number analyzed (Scores on a Scale) | 100 | 100
Scores on a VAS Scale | 44.9 (31.5) | 14.7 (17.7)

2. Secondary Outcome: Wrinkle Improvement at Day 14
Description: This measure was performed by the validated GAIS tool (Global Asthetic Improvement Scale). The GAIS was completed by the participant at day 14. The GAIS is a qualitative 5 point scale evaluating Aesthetic Improvement (0=worse, 1=no change, 2=Improved, 3=Much Improved, 4=very much improved). Treatment success is defined as at least a one grade improvement (2, 3, or 4) from pre-treatment.
Time Frame: 14 days after treatment when compared to baseline
Measure: Number; unit: participants
Groups:
- Restylane-L Side of Face: Restylane with Lidocaine gel(Restylane-L) side of the face. Injection occurs on Day 1 only. Injection amount is determined by achieving the optimal cosmetic results (variable).
- Restylane Side of Face: The Restylane gel side of the face. Injection occurs on Day 1 only. Injection amount is determined by achieving the optimal cosmetic results (variable).
Arm/Group | Restylane-L Side of Face | Restylane Side of Face
Number analyzed (Participants) | 60 | 60
participants | 60 | 59

ADVERSE EVENTS:
Arm/Group | Restylane-L Side of Face | Restylane Side of Face
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 46/60 | 46/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane-L Side of Face (N=60) | Restylane Side of Face (N=60)
Ecchymosis (Vascular disorders) | 23 (23) | 19 (19)
Edema (General disorders) | 24 (24) | 22 (22)
Erythema (General disorders) | 28 (28) | 27 (27)
Tenderness (General disorders) | 23 (23) | 26 (26)
Pain (General disorders) | 17 (17) | 18 (18)
Pruitis (General disorders) | 6 (6) | 4 (4)
Papule (General disorders) | 1 (1) | 2 (2)
Vasospasm (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less